CLINICAL TRIAL: NCT00823121
Title: Can Fresh Embryo Transfers be Replaced by Cryopreserved-thawed Embryo Transfers in Assisted Reproductive Cycles?
Brief Title: Replacement of Fresh Embryo Transfers (ETs) by Frozen Embryo Transfers (FETs) Using Vitrification
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yazd Research & Clinical Center for Infertility (Other)
Responsible Party: abbas,aflatoonian, YazdRCCI
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 654YazdRCCI
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2009-04

CONDITIONS: In Vitro Fertilization
Keywords: Fresh embryo transfer; frozen- thawed embryo transfer; vitrification; endometrial receptivity; implantation rate; pregnancy; ART
MeSH Terms: interventions — Buserelin; follitropin alfa; Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- frozen-embryo transfer (Active Comparator): In this group all embryos are cryopreserved and two months later embryo transfer will perform.
  Interventions: Procedure: freezing embryos by vitrification; Drug: buserelin; Drug: recombinant FSH; Drug: human chorionic gonadotropin (pregnyl)
- fresh embryo transfer (Active Comparator): In this arm fresh embryo transfers are performed on day 2 or 3.
  Interventions: Procedure: fresh embryo transfers; Drug: buserelin; Drug: recombinant FSH; Drug: human chorionic gonadotropin (pregnyl)

INTERVENTIONS:
Procedure: freezing embryos by vitrification — vitrification by Cryotop method
  Other Names: cryopreservation of embryos
  Arms: frozen-embryo transfer
Procedure: fresh embryo transfers — fresh embryo transfers
  Other Names: embryo transfer using fresh embryos
  Arms: fresh embryo transfer
Drug: buserelin — Daily administration of 500 µg subcutaneous buserelin from day 21 of menstrual cycle; reduce to 250 µg daily when ovarian suppression is confirmed.
  Other Names: suprefact
Drug: recombinant FSH — gonadotropin stimulation with rFSH 150 IU/day from day 2 of menstrual cycle
  Other Names: Gonal F
Drug: human chorionic gonadotropin (pregnyl) — hCG 10,000 IU is administered when at least 2 follicles reach a mean diameter of 18 mm.
  Other Names: pregnyl

SUMMARY:
Cryopreservation of all embryos and transferring them subsequently in assisted reproductive technology (ART) cycles to improve outcome.

DETAILED DESCRIPTION:
All patients in the initial cohort were treated with long protocol for ovarian stimulation. For pituitary down-regulation, patients were treated with daily administration of 0.5 mg buserelin (suprefact, Aventis, Frankfurt, Germany) from day 21 of menstrual cycle. Buserelin was reduced to 0.25 mg daily when ovaries were quiescent on ultrasound, and COH was initiated with recombinant FSH (Gonal F, Serono, Aubnne, Switzerland) 150 IU/day on day 2 of withdrawal bleeding. Serial ultrasound examinations and evaluation of serum E2 levels were used to assess ovarian response, and then gonadotropin dose adjustments were done as required. Human chorionic gonadotropin (pregnyl, Organon, Oss, the Netherlands ) 10,000 IU was administered when at least two follicles reached a mean diameter of 18 mm.

Oocyte retrieval was performed 34-36 hours after hCG administration and conventional insemination or ICSI was performed as clinically appropriate.

In 187 patients allocated to fresh ET group, ET were performed on the day 2. Embryos were transferred under ultrasound guidance, with a C.C.D. embryo transfer catheter (Laboratory C.C.D., Paris, France). Luteal support with progesterone in oil (Progesterone, Aburaihan Co., Tehran, Iran) 100 mg daily IM was started on the day of oocyte retrieval and continued until the documentation of fetal heart activity on ultrasound.

In 187 patients allocated to FET group, cryopreservation of all embryos were undertaken with vitrification by Cryotop method and after two months, embryos were transferred.

The protocol for the Cryotop vitrification of embryos was described previously (Kuwayama et al., 2005; Kuwayama, 2007).

After a two-step loading with equilibration solution containing 7.5% (v/v) ethylene glycol and 7.5% (v/v) dimethyl sulfoxide, and vitrification solution containing 15% (v/v) ethylene glycol, 15% (v/v) dimethyl sulfoxide and 0.5 mol/L sucrose, embryos were loaded with a narrow glass capillary onto the Cryotop in a volume of < 0.1 µL . After loading, almost all the solution was removed to leave only a thin layer covering the embryos, and the sample was quickly immersed into liquid nitrogen (LN). Subsequently, the plastic cap was pulled over the film part of the Cryotop, and the sample was stored under LN. At warming, the protective cap was removed from the Cryotop while it was still submerged in LN and the Cryotop was immersed directly into a 37˚C medium containing sucrose. The embryos were then sequentially incubated in diluents solution before further in vitro culture for transfer.

Patients were prepared for ET with oral E2 to attain endometrial thickness ≥ 8 mm and triple line pattern on ultrasound scans. At that time, patients were given 100 mg of IM progesterone in oil daily and ET was preformed three days later under abdominal ultrasound guidance as described earlier. Oral E2 and progesterone were continued until documentation of fetal heart activity by ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* age < 38
* normal day 3 FSH
* classified as high risk for OHSS
* has ≥ 15 follicles with a mean diameter ≥ 12 mm per each ovary
* E2 levels on the day of hCG administration > 3000 pg/mL
* undergoing her first assisted reproduction treatment cycle

Exclusion Criteria:

* who does not have good-quality embryos appropriate for cryopreservation

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-02 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
implantation rate | 4 weeks

SECONDARY OUTCOMES:
on going pregnancy rate | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: abbas aflatoonian, M.D., Principal Investigator — Research and Clinical Center for Infertility; homa oskouian, M.D., Principal Investigator — Research and Clinical Center for Infertility
Locations (1):
- : Research and clinical center for infertility, Yazd, Yazd Province, Iran

REFERENCES:
- [Derived] Aflatoonian A, Oskouian H, Ahmadi S, Oskouian L. Can fresh embryo transfers be replaced by cryopreserved-thawed embryo transfers in assisted reproductive cycles? A randomized controlled trial. J Assist Reprod Genet. 2010 Jul;27(7):357-63. doi: 10.1007/s10815-010-9412-9. Epub 2010 Apr 6. PMID 20373015 (Retraction: PMID 23975193 J Assist Reprod Genet. 2013 Sep;30(9):1245)